CLINICAL TRIAL: NCT06569693
Title: Dyadic Sleep Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Youngmee Kim, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20240214; R21NR021083 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSOS Intervention Group (Experimental): Participants (patient-sleep-partner caregiver dyads) in this group will receive the My Sleep Our Sleep (MSOS) intervention. Total participation is up to 13 weeks.
  Interventions: Behavioral: My Sleep Our Sleep (MSOS) Program
- BBTI Intervention Group (Experimental): Participants (patient-sleep-partner caregiver dyads) in this group will receive the Brief Behavioral Treatment for Insomnia (BBTI). Total participation is up to 13 weeks.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia (BBTI)

INTERVENTIONS:
Behavioral: My Sleep Our Sleep (MSOS) Program — MSOS is a sleep intervention developed by the investigator aimed at improving sleep health for patient-sleep-partner caregiver dyads using behavioral education in sleep behaviors, sleep cognition and sleep in relationship.
  MSOS will be delivered over four weeks, in weekly one-hour sessions, one session per week.
  Other Names: MSOS
  Arms: MSOS Intervention Group
Behavioral: Brief Behavioral Treatment for Insomnia (BBTI) — BBTI is brief patient-focused intervention for patient-sleep-partner caregiver dyads, aimed at altering participants' sleep behaviors to improve sleep. BBTI utilizes behavioral education in sleep restriction and stimulus control. For sleep restriction, participants will be instructed to limit the time they spend in bed, which serves to increase sleep efficiency. For stimulus control, participants will be instructed to go to bed only when feeling sleepy and reserve the bed for sleep and intimacy.
  BBTI will be delivered over four weeks, in weekly one-hour sessions, one session per week.
  Other Names: BBTI
  Arms: BBTI Intervention Group

SUMMARY:
The purpose of this study is to learn about sleep behaviors and test different ways to help patients with cancer and caregiver partners.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria for patients are:

  * newly diagnosed with stage I to IV of a GI cancer (anus, colon, esophagus, gallbladder, large and small intestine, liver, pancreas, rectum, stomach, other biliary or digestive organs)
  * diagnosis in the past 12 months at the time of enrollment
  * having a consistent sleep partner.
* The eligibility criterion for caregivers is:

  * a sleep partner of the patient.
* Additional eligibility criteria for both patients and caregivers are:

  * Pittsburgh Sleep Quality Index (PSQI) ≥ 5,
  * willing to change sub-optimal sleep habits,
  * 18 years or older,
  * able to speak/listen English at the 8th grade level for intervention sessions,
  * able to read English or Spanish at the 8th grade for self-reported questionnaires,
  * > 4 weeks after surgery, if any, prior to enrollment, and no surgery planned in the next 5 weeks during the study period because surgery affects sleep.

Exclusion Criteria:

* Exclusion criteria for both patients and caregivers are having had a diagnosis of major depressive disorder, psychosis, or bipolar disorder that is not currently treated;
* Active suicidality, or substance or alcohol dependency in the past year;
* Currently have narcolepsy, restless leg syndrome, or untreated sleep apnea that is screened using the Sleep Health Screen;
* Both patients and caregivers have an extreme chronotype, or do shift work to have no overlap in sleep schedule between them; and plan trans-meridian travel during the period of data collection blocks; and having hearing or visual impairment, dementia, or cognitive dysfunction.
* Adults unable to consent, individuals who are not yet adults, pregnant women, or prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in sleep disturbance symptoms as measured by scores on the Pittsburgh Sleep Quality Index (PSQI) | Baseline, Up to 13 weeks
  Change in sleep disturbance symptoms (patient-sleep-partner caregiver dyads) among participants will be compared and reported for both intervention groups, BBTI and MSOS, as measured by scores on the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-reported, 19-item questionnaire health-related quality of life (HRQOL) questionnaire which assesses sleep quality and disturbances at baseline, week 5 and week 13. Questions generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. A decrease of ≥ 5 points on the PSQI) will be considered as clinical improvement of symptoms.

SECONDARY OUTCOMES:
Change in insomnia symptoms as measured by scores on the Insomnia Severity Index (ISI) | Baseline, Up to 13 weeks
  Change in insomnia symptoms among participants (patient-sleep-partner caregiver dyads) will be compared and reported for both intervention groups, BBTI and MSOS, as measured by scores on the 7-item Insomnia Severity Index (ISI). The ISI is a self-reported, health-related quality of life (HRQOL) questionnaire used to assess insomnia symptoms at baseline, week 5 and week 13. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, notice ability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item, ranging from 0 to 4 (e.g., 0 = no problem; 4 = very severe problem). The total score ranges from 0 to 28, the lower total score indicates a lower level of insomnia. Greater than a 6-point decrease on the ISI is considered substantial reduction in insomnia symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Youngmee Kim, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Tsai TC, Steel JL, Ramos AR, Laurenceau JP, Troxel WM. Protocol of testing the feasibility and acceptability of two brief dyadic sleep interventions for adults with cancer and their bedpartner caregivers. Pilot Feasibility Stud. 2025 Jun 14;11(1):82. doi: 10.1186/s40814-025-01671-z. PMID 40514758